CLINICAL TRIAL: NCT00221364
Title: Trachoma Elimination With Repeated Mass Azithromycin Treatments
Brief Title: Trachoma Elimination Follow-up
Acronym: TEF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 10-02630
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Trachoma; Chlamydia
Keywords: Trachoma; Chlamydia; Azithromycin
MeSH Terms: conditions — Trachoma; Chlamydia Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Mass treatment with oral azithromycin to an entire village

SUMMARY:
The WHO has initiated a program to eliminate blinding trachoma by the year 2020, in large part by mass oral azithromycin distributions. It is not clear how frequently or for how long these treatments are necessary. Here we assess the frequency and duration of treatment.

DETAILED DESCRIPTION:
40 villages in the Gurage Zone of Ethiopia were randomly assigned to biannual treatment, annual treatment, and a single treatment. Each treatment consisted of a single dose of oral azithromycin to the entire population over the age of 1 year (when the study was started, azithromycin had not yet been approved for ages below 1 year). We assess the prevalence the ocular chlamydia that causes trachoma in the peak prevalence age of 1-5 years at baseline, and 2, 6, 12, 18, and 24 months post treatment. An extension of the study monitors infection at 30 and 36 months post treatment. Untreated villages from the same area are enrolled in a step-wedge design to assess the presence of a secular trend. A random sample of those not within the 1-5 year old age group are examined to assess the prevalence of infection in the entire community.

ELIGIBILITY:
Inclusion Criteria:

Age 1 to 5 years old in a village in the Gurage zone with endemic trachoma

Exclusion Criteria:

Refusal of village chief (for village inclusion), or refusal of parent or guardian (for individual inclusion)

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 2003-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
The prevalence of ocular chlamydia infection in a village as determined by PCR

SECONDARY OUTCOMES:
Clinical active trachoma, as determined by the WHO simplified grading system, by village

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Lietman, MD, Principal Investigator — Proctor Foundation, UCSF
Locations (1):
- ORBIS-Ethiopia, Addis Ababa, Ethiopia

REFERENCES:
- [Background] Melese M, Chidambaram JD, Alemayehu W, Lee DC, Yi EH, Cevallos V, Zhou Z, Donnellan C, Saidel M, Whitcher JP, Gaynor BD, Lietman TM. Feasibility of eliminating ocular Chlamydia trachomatis with repeat mass antibiotic treatments. JAMA. 2004 Aug 11;292(6):721-5. doi: 10.1001/jama.292.6.721. PMID 15304470
- [Background] Chidambaram JD, Melese M, Alemayehu W, Yi E, Prabriputaloong T, Lee DC, Cevallos V, Zhou Z, Whitcher JP, Gaynor BD, Lietman TM. Mass antibiotic treatment and community protection in trachoma control programs. Clin Infect Dis. 2004 Nov 1;39(9):e95-7. doi: 10.1086/424747. Epub 2004 Oct 6. PMID 15494901
- [Background] Ray KJ, Porco TC, Hong KC, Lee DC, Alemayehu W, Melese M, Lakew T, Yi E, House J, Chidambaram JD, Whitcher JP, Gaynor BD, Lietman TM. A rationale for continuing mass antibiotic distributions for trachoma. BMC Infect Dis. 2007 Aug 7;7:91. doi: 10.1186/1471-2334-7-91. PMID 17683646
- [Background] Lee S, Alemayehu W, Melese M, Lakew T, Lee D, Yi E, Cevallos V, Donnellan C, Zhou Z, Chidambaram JD, Gaynor BD, Whitcher JP, Lietman TM. Chlamydia on children and flies after mass antibiotic treatment for trachoma. Am J Trop Med Hyg. 2007 Jan;76(1):129-31. PMID 17255240
- [Background] Chidambaram JD, Alemayehu W, Melese M, Lakew T, Yi E, House J, Cevallos V, Zhou Z, Maxey K, Lee DC, Shapiro BL, Srinivasan M, Porco T, Whitcher JP, Gaynor BD, Lietman TM. Effect of a single mass antibiotic distribution on the prevalence of infectious trachoma. JAMA. 2006 Mar 8;295(10):1142-6. doi: 10.1001/jama.295.10.1142. PMID 16522834
- [Background] Haug S, Lakew T, Habtemariam G, Alemayehu W, Cevallos V, Zhou Z, House J, Ray K, Porco T, Rutar T, Keenan J, Lietman TM, Gaynor BD. The decline of pneumococcal resistance after cessation of mass antibiotic distributions for trachoma. Clin Infect Dis. 2010 Sep 1;51(5):571-4. doi: 10.1086/655697. PMID 20649409
- [Background] Shah NA, House J, Lakew T, Alemayehu W, Halfpenny C, Hong KC, Keenan JD, Porco TC, Whitcher JP, Lietman TM, Gaynor BD. Travel and implications for the elimination of trachoma in ethiopia. Ophthalmic Epidemiol. 2010 Mar;17(2):113-7. doi: 10.3109/09286581003624921. PMID 20302432
- [Background] Keenan JD, Lakew T, Alemayehu W, Melese M, Porco TC, Yi E, House JI, Zhou Z, Ray KJ, Acharya NR, Whitcher JP, Gaynor BD, Lietman TM. Clinical activity and polymerase chain reaction evidence of chlamydial infection after repeated mass antibiotic treatments for trachoma. Am J Trop Med Hyg. 2010 Mar;82(3):482-7. doi: 10.4269/ajtmh.2010.09-0315. PMID 20207878
- [Background] Biebesheimer JB, House J, Hong KC, Lakew T, Alemayehu W, Zhou Z, Moncada J, Roger A, Keenan J, Gaynor BD, Schachter J, Lietman TM. Complete local elimination of infectious trachoma from severely affected communities after six biannual mass azithromycin distributions. Ophthalmology. 2009 Nov;116(11):2047-50. doi: 10.1016/j.ophtha.2009.04.041. Epub 2009 Sep 10. PMID 19744717
- [Background] Lakew T, Alemayehu W, Melese M, Yi E, House JI, Hong KC, Zhou Z, Ray KJ, Porco TC, Gaynor BD, Lietman TM, Keenan JD. Importance of coverage and endemicity on the return of infectious trachoma after a single mass antibiotic distribution. PLoS Negl Trop Dis. 2009 Aug 25;3(8):e507. doi: 10.1371/journal.pntd.0000507. PMID 19707573
- [Background] Lakew T, House J, Hong KC, Yi E, Alemayehu W, Melese M, Zhou Z, Ray K, Chin S, Romero E, Keenan J, Whitcher JP, Gaynor BD, Lietman TM. Reduction and return of infectious trachoma in severely affected communities in Ethiopia. PLoS Negl Trop Dis. 2009;3(2):e376. doi: 10.1371/journal.pntd.0000376. Epub 2009 Feb 3. PMID 19190781
- [Background] Hong KC, Schachter J, Moncada J, Zhou Z, House J, Lietman TM. Lack of macrolide resistance in Chlamydia trachomatis after mass azithromycin distributions for trachoma. Emerg Infect Dis. 2009 Jul;15(7):1088-90. doi: 10.3201/eid1507.081563. PMID 19624926
- [Background] Yang JL, Hong KC, Schachter J, Moncada J, Lekew T, House JI, Zhou Z, Neuwelt MD, Rutar T, Halfpenny C, Shah N, Whitcher JP, Lietman TM. Detection of Chlamydia trachomatis ocular infection in trachoma-endemic communities by rRNA amplification. Invest Ophthalmol Vis Sci. 2009 Jan;50(1):90-4. doi: 10.1167/iovs.08-2247. Epub 2008 Aug 8. PMID 18689701
- [Background] Melese M, Alemayehu W, Lakew T, Yi E, House J, Chidambaram JD, Zhou Z, Cevallos V, Ray K, Hong KC, Porco TC, Phan I, Zaidi A, Gaynor BD, Whitcher JP, Lietman TM. Comparison of annual and biannual mass antibiotic administration for elimination of infectious trachoma. JAMA. 2008 Feb 20;299(7):778-84. doi: 10.1001/jama.299.7.778. PMID 18285589
- [Background] Gill DA, Lakew T, Alemayehu W, Melese M, Zhou Z, House JI, Hong KC, Ray KJ, Gandhi N, Whitcher JP, Gaynor BD, Lietman TM. Complete elimination is a difficult goal for trachoma programs in severely affected communities. Clin Infect Dis. 2008 Feb 15;46(4):564-6. doi: 10.1086/526777. PMID 18194094
- [Background] Keenan JD, Lakew T, Alemayehu W, Melese M, House JI, Acharya NR, Porco TC, Gaynor BD, Lietman TM. Slow resolution of clinically active trachoma following successful mass antibiotic treatments. Arch Ophthalmol. 2011 Apr;129(4):512-3. doi: 10.1001/archophthalmol.2011.46. No abstract available. PMID 21482879
- [Derived] Cevallos V, Whitcher JP, Melese M, Alemayehu W, Yi E, Chidambaram JD, Lee S, Reddy H, Gaynor BD, Lietman TM, Keenan JD. Association of conjunctival bacterial infection and female sex in cicatricial trachoma. Invest Ophthalmol Vis Sci. 2012 Aug 7;53(9):5208-12. doi: 10.1167/iovs.12-9984. PMID 22736616
- [Derived] See CW, Alemayehu W, Melese M, Zhou Z, Porco TC, Shiboski S, Gaynor BD, Eng J, Keenan JD, Lietman TM. How reliable are tests for trachoma?--a latent class approach. Invest Ophthalmol Vis Sci. 2011 Aug 3;52(9):6133-7. doi: 10.1167/iovs.11-7419. PMID 21685340